CLINICAL TRIAL: NCT00668096
Title: A Randomized, Double Blind, Placebo Controlled, Flexible Dose, Multicentre Study of Levitra in a Broad Population of Men With Erectile Dysfunction and Previously Untreated With PDE5 Inhibitors.
Brief Title: A Randomised Study of Levitra to Treat Men With Erections Problems and Previously Untreated With Similar Therapy.
Acronym: FINDER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11334
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Last update posted 2014-12-25 (Estimated); Status verified 2014-12

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction; PDE5 inhibitors
MeSH Terms: conditions — Erectile Dysfunction | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo
- Arm 1 (Experimental)
  Interventions: Drug: Levitra (Vardenafil, BAY38-9456)

INTERVENTIONS:
Drug: Levitra (Vardenafil, BAY38-9456) — Vardenafil 5 mg or 10 mg or 20 mg, orally1 hour prior to sexual activity
  Arms: Arm 1
Drug: Placebo — Matching Placebo
  Arms: Arm 2

SUMMARY:
The objective of this study was to evaluate the efficacy and tolerability of the phosphodiesterase type 5 inhibitor (PDE5 inhibitor), vardenafil, in a broad population of subjects with erectile dysfunction of different aetiologies and severity, who have not been previously treated with a PDE5 inhibitor; Efficacy and safety was compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Males with erectile dysfunction according to the National Institute of Health (NIH) Consensus statement (inability to attain and/or maintain penile erection sufficient for satisfactory sexual performance
* Heterosexual relationship for more than 6 months
* Partner willing to complete the TSS

Exclusion Criteria:

* Primary hypoactive sexual desire
* History of myocardial infarction, stroke or life-threatening arrhythmia within the prior 6 months
* Nitrate use
* Other exclusion criteria apply according to the Summary of Product Characteristics

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 260 (Actual)
Dates: Start 2004-05; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Hierarchical significance testing was applied to the 3 primary efficacy parameters at the 5% significance level. Parameters were to be tested: GAQ first, Sexual Encounter Profile 3 second and SEP 2 third. SEP 3 will only be tested if GAQ is sign. | 16 weeks

SECONDARY OUTCOMES:
International Index of Erectile Function | 16 weeks
Treatment Satisfaction Scale | 16 weeks
Other patient diary based variables | 16 weeks
Safety and tolerability | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (33):
- Belgium (4):
  - Bruxelles - Brussel
  - Drieslinter
  - Genk
  - Leuven
- Denmark (4):
  - Gentofte Municipality
  - Næstved
  - Svendborg
  - Viborg
- Finland (3):
  - Kerava
  - Oulu
  - Tampere
- France (5):
  - Grenoble
  - Lille
  - Lyon
  - Marseille
  - Montpellier
- Germany (9):
  - Hamburg, Hamburg
  - Dresden, Saxony
  - Leipzig, Saxony
  - Leisnig, Saxony
  - Meissen, Saxony
  - Harrislee, Schleswig-Holstein
  - Norderstedt, Schleswig-Holstein
  - Wahlstedt, Schleswig-Holstein
  - Altenburg, Thuringia
- Spain (4):
  - Barcelona, Barcelona
  - Gavà, Barcelona
  - L'Hospitalet de Llobregat, Barcelona
  - Badalona (Barcelona), Catalonia
- United Kingdom (4):
  - Crowborough, East Sussex
  - Chipping Norton, Oxfordshire
  - Lichfield, Staffordshire
  - Hamilton, Strathclyde